CLINICAL TRIAL: NCT05782790
Title: Development of Action Observation Therapy Program in Patients With Neurogenic Dysphagia and Investigation of Its Efficacy
Brief Title: Action Observation Therapy Program in Patients With Neurogenic Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ARZUCAN TOKSAL, Lecturer, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: ZBEU
Record Dates: First submitted 2023-03-07; First posted 2023-03-24 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Neurogenic Dysphagia; Rehabilitation; Deglutition Disorders
Keywords: Neurogenic Dysphagia; Rehabilitation
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Observation Therapy Group (Experimental): In this method, patients will be seated in a comfortable chair in front of a 32-inch television placed approximately 2 meters away in a quiet room. On television, videos that will be used in swallowing rehabilitation prepared on realistic animations and/or real models will be shown to the patients. Patients will be asked to watch these exercise videos for 20 minutes with their full attention and concentrate on how the actions are done. Patients; While watching the videos, they will not be asked to do any movement, they will be asked to imitate the exercises after the videos are finished.
  Interventions: Behavioral: Action Observation Theraphy Group
- Classic Swallowing Exercise Group (Experimental): Exercises include positioning, swallowing maneuvers, food modification, and swallowing exercises, which are sensory stimulation, oral motor exercises, head-neck mobilization, Shaker exercises, and neck region and tongue strengthening exercises, which are compensatory strategies according to the swallowing rehabilitation program accepted in the literature.
  Interventions: Behavioral: Classic Swallowing Exercise Group

INTERVENTIONS:
Behavioral: Action Observation Theraphy Group — In this method, patients will be seated in a comfortable chair in front of a 32-inch television placed approximately 2 meters away in a quiet room. On television, videos that will be used in swallowing rehabilitation prepared on realistic animations and/or real models will be shown to the patients. Patients will be asked to watch these exercise videos for 20 minutes with their full attention and concentrate on how the actions are done.
  Evaluations to be made before starting the treatment program and finished; demographic information, Standardized Mini Mental Test, Turkish Eating Assessment Tool, Videofluoroscopic Swallowing Study (VFYC), Penetration Aspiration Scale (PAS), Evaluation of Swallowing Ability and Function, Surface Electromyographic Measurements of Suprahyoid Muscles, Swallowing Quality of Life Questionnaire, Beck Depression Scale.
  Arms: Action Observation Therapy Group
Behavioral: Classic Swallowing Exercise Group — Exercises include positioning, swallowing maneuvers, food modification, and swallowing exercises, which are sensory stimulation, oral motor exercises, head-neck mobilization, Shaker exercises, and neck region and tongue strengthening exercises, which are compensatory strategies according to the swallowing rehabilitation program accepted in the literature. Evaluations to be made before starting the treatment program and finished; demographic information, Standardized Mini Mental Test, Turkish Eating Assessment Tool, Videofluoroscopic Swallowing Study (VFYC), Penetration Aspiration Scale (PAS), Evaluation of Swallowing Ability and Function, Surface Electromyographic Measurements of Suprahyoid Muscles, Swallowing Quality of Life Questionnaire, Beck Depression Scale.
  Arms: Classic Swallowing Exercise Group

SUMMARY:
Swallowing is the delivery of food taken from the mouth to the stomach at an appropriate rate with the sequential movements of the structures in the oral, pharyngeal, and esophageal regions. The change in swallowing function due to structural and functional changes in the structures responsible for swallowing is called swallowing disorder (dysphagia). The treatment of neurogenic dysphagia aims to prevent complications such as dysphagia-related aspiration pneumonia, airway obstructions, and malnutrition, and to regulate swallowing physiology. Swallowing rehabilitation created for this purpose consists of compensatory techniques and rehabilitation methods. Compensatory techniques include changing the consistency and properties of food, postural changes, and increasing voluntary control. Rehabilitation methods consist of exercise-based methods such as oral motor exercises, Shaker exercises, and tongue strengthening exercises. In addition to these rehabilitation methods, it has been reported that neuromuscular electrical stimulation (NMES) positively affects swallowing function. It is known that cortical reorganization occurs due to sensory restimulation following the exercises performed in dysphagia rehabilitation. It has been reported that swallowing rehabilitation may also have positive effects on neural plasticity in patients with dysphagia. It is essential to transfer approaches that support neural plasticity to swallowing rehabilitation. The starting point of action observation therapy (AOT), which has just entered the literature, is based on motor learning-based approaches used in neurological rehabilitation, neural plasticity, motor imagery, and mirror neurons. Based on the fact that both motor image and movement observation can play a role in (re)learning motor control, AOT aims to provide activation of motor areas with movement observation and to develop a rehabilitation approach based on performing the observed actions. The AOT method consists of two stages. First, videos of the exercises to be done are created, and in the first stage, patients are asked to watch the video by focusing only on the video. In the second stage, patients need to practice the exercises they follow themselves. In this way, it is thought that the effectiveness of both motor learning will be increased. When studies on patients with neurogenic dysphagia are examined, the use of AOT, which is a new approach, in swallowing rehabilitation has not been found. Therefore, in this study, the creation of an AOT program based on mirror neuron and motor learning theory and its effect on swallowing function and quality of life related to swallowing will be examined in patients with neurogenic dysphagia. The investigators aim to increase the healing efficiency of the AOT program in patients with neurogenic dysphagia.

DETAILED DESCRIPTION:
The treatment of neurogenic dysphagia aims to prevent complications such as dysphagia-related aspiration pneumonia, airway obstructions, and malnutrition, and to regulate swallowing physiology. Swallowing rehabilitation created for this purpose consists of compensatory techniques and rehabilitation methods. Compensatory techniques include changing the consistency and properties of food, postural changes, and increasing voluntary control. Rehabilitation methods consist of exercise-based methods such as oral motor exercises, Shaker exercises, and tongue strengthening exercises. In addition to these rehabilitation methods, it has been reported that neuromuscular electrical stimulation (NMES) positively affects swallowing function. It is known that cortical reorganization occurs due to sensory restimulation following the exercises performed in dysphagia rehabilitation. It has been reported that swallowing rehabilitation may also have positive effects on neural plasticity in patients with dysphagia. It is essential to transfer approaches that support neural plasticity to swallowing rehabilitation. The starting point of action observation therapy (AOT), which has just entered the literature, is based on motor learning-based approaches used in neurological rehabilitation, neural plasticity, motor imagery, and mirror neurons. Based on the fact that both motor image and movement observation can play a role in (re)learning motor control, AOT aims to provide activation of motor areas with movement observation and to develop a rehabilitation approach based on performing the observed actions. The AOT method consists of two stages. First, videos of the exercises to be done are created, and in the first stage, patients are asked to watch the video by focusing only on the video. In the second stage, patients need to practice the exercises they follow themselves. In this way, it is thought that the effectiveness of both motor learning will be increased. When studies on patients with neurogenic dysphagia are examined, the use of AOT, which is a new approach, in swallowing rehabilitation has not been found. Therefore, in this study, the creation of a AOT program based on mirror neuron and motor learning theory and its effect on swallowing function and quality of life-related to swallowing will be examined in patients with neurogenic dysphagia. The investigators aim to increase the healing efficiency of the AOT program in patients with neurogenic dysphagia.

A Videofluoroscopic Swallowing Study was performed in the Zonguldak Bülent Ecevit University Department of Radiology, routinely directed by the relevant neurologist, with any neurological disease over the age of 18, who applied to the Zonguldak Bülent Ecevit University Neurology Outpatient Clinic, and as a result, Penetration Aspiration Score score of 2 and above was performed. Individuals with a Standardized Mini-Mental Test score of 24 and above will be included voluntarily.

After the individuals included in the study have read and accepted the informed consent form, the following evaluations will be applied first. According to the sample selection criteria, the patients included in the study will be randomly divided into two groups the observational movement therapy group and the classical swallowing exercises group. Swallowing rehabilitation including appropriate exercises specific to the clinical conditions of the patients will be created. While these exercises are given to the observational movement therapy group with the AOT program, the patients in the classical swallowing exercises group will practice without watching the video. The following evaluations will be made to the patients before starting the exercise sessions and after the 4-week exercise sessions are over.

Evaluations to be made before starting the treatment program; demographic information, Standardized Mini Mental Test, Turkish Eating Assessment Tool, Videofluoroscopic Swallowing Study (VFYC), Penetration Aspiration Scale (PAS), Evaluation of Swallowing Ability and Function, Surface Electromyographic Measurements of Suprahyoid Muscles, Swallowing Quality of Life Questionnaire, Beck Depression Scale.

Evaluations to be made after the treatment program; Turkish Eating Assessment Tool, Evaluation of Swallowing Ability and Function, Superficial Electromyographic Measurements of Suprahyoid Muscles, Swallowing Quality of Life Questionnaire (SWAL-QOL), Beck Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Having a neurological diagnosis
* Having been directed by a neurologist for the diagnosis of dysphagia, performed VFYC in the Department of Radiology, and having a Penetration Aspiration Scale score of 2 or higher as a result of VFYC
* Standardized Mini Mental Test score of 24 or higher

Exclusion Criteria:

* Receiving swallowing rehabilitation before
* Head and neck surgery deliveries and a history of other diseases involving swallowing difficulties
* Individuals with tracheostomy
* Any vision or hearing problems
* Cognitive status results from any other infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Surface Electromyographic Measurements of the Suprahyoid Muscles | 2 years
  yEMG, which provides practical objective data and provides electrical activation information directly from the relevant muscles, will measure the activation development in the muscles during the maximum voluntary isometric contractions to be made during a standard activity (drinking 10 ml of water). The EMG measurement to be applied to the participants will be done outside working hours in a way that will not disrupt routine patient functioning. The electrodes to be used in EMG will be covered by the researchers. This assessment will be applied before the start of the exercise program and at the end of the exercise program at the end of the 4th week.

SECONDARY OUTCOMES:
Turkish Version of the Eating Assessment Tool-10 - T-EAT-10 | 2 years
  The Eating Assessment Tool is a valid and reliable outcome measure that includes symptom-specific questions about own swallowing function. The Turkish version, validity, and reliability study was conducted in 2016. T-EAT-10 is an easy and quick swallowing difficulty screening test consisting of 10 questions. The patient scores each question from 0 (no problem) to 4 (serious problem). The total score is obtained by adding the scores given to each item. The minimum score is 0, the maximum score is 40. High scores indicate a swallowing disorder. A total of 3 points or more is significant in terms of swallowing disorder risk. A high score indicates a symptom of excessive swallowing disorder.
Swallowing Ability and Function Evaluation-SAFE | 2 years
  This scale used to evaluate swallowing function is SAFE. swallowing function; The oropharyngeal mechanism and physical examination, oral phase swallowing assessment, and pharyngeal phase swallowing assessment include a three-stage assessment. In the oropharyngeal mechanism and physical examination step, lips, tongue, palate, cheeks, teeth, jaw, larynx functions, and oral reflex are observed, and at the end of this step, the physical examination (FM) total score is obtained. The total score will be calculated out of 30 and the higher the score, the worse the swallowing function.
Swallowing Quality of Life questionnaire (SWAL-QOL) | 2 years
  SWAL-QOL evaluates the impact of swallowing disorder on quality of life from patient sources. It consists of 44 questions evaluating different dimensions of quality of life. Each question is scored from 1 to 5 (1: completely true, 5: not at all true). It has been reported that as the score increases, the quality of life-related to swallowing worsens. It has 11 subheadings: general complaints, desire to eat, time to eat, social, food choice, fear of eating, sleep, fatigue, communication, mental health, and symptom frequency. The Turkish validity and reliability of this questionnaire, which evaluates the quality of life due to swallowing, was performed. This questionnaire will be used in this study to evaluate the patient's quality of life-related to swallowing.
Beck Depression Scale | 2 years
  Developed by Aaron T. Beck and studied in Turkish version, 21 multiple-choice questions is a tool used to measure the severity of depression. Its scoring ranges from 0 to 63; A score of 0-9 indicates minimal depressive symptoms, 10-16 points indicates mild depressive symptoms, 17-29 points indicates moderate depressive symptoms, and 30-63 points indicates severe depressive symptoms. Since the Beck Depression Scale is a comprehensive questionnaire that measures the symptoms of depression in the human body and its mental state, it will be used in our study to measure the severity of depression in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Bilgin, Prof, Study Director — Hacettepe University
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panebianco M, Marchese-Ragona R, Masiero S, Restivo DA. Dysphagia in neurological diseases: a literature review. Neurol Sci. 2020 Nov;41(11):3067-3073. doi: 10.1007/s10072-020-04495-2. Epub 2020 Jun 7. PMID 32506360
- [Background] Rocca MA, Meani A, Fumagalli S, Pagani E, Gatti R, Martinelli-Boneschi F, Esposito F, Preziosa P, Cordani C, Comi G, Filippi M. Functional and structural plasticity following action observation training in multiple sclerosis. Mult Scler. 2019 Oct;25(11):1472-1487. doi: 10.1177/1352458518792771. Epub 2018 Aug 7. PMID 30084706
- [Derived] Toksal Ucar A, Piri Cinar B, Alicioglu B, Bostan G, Bilgin S. Application of Action Observation Therapy in Swallowing Rehabilitation: A Randomised Controlled Study. J Oral Rehabil. 2025 Mar;52(3):320-331. doi: 10.1111/joor.13902. Epub 2024 Nov 26. PMID 39599964